CLINICAL TRIAL: NCT06336863
Title: An Extension Protocol for Subjects Previously Enrolled in the "Use of Donor Derived-cell Free DNA (AlloSure) and Gene Expression Profiling (AlloMap Kidney) to Facilitate Belatacept Monotherapy in Kidney Transplant Patients"
Brief Title: Use of DNA Testing and Gene Expression Profiling to Help Transition Kidney Transplant Recipients to Belatacept-only Immunosuppression
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, David Wojciechowski, Associate Professor, Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-1151
Record Dates: First submitted 2024-03-21; First posted 2024-03-29 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Kidney Transplant Immunosuppression
Keywords: Belatacept Monotherapy; Kidney Transplant Recipients; Immunosuppression; Weaning; DNA Testing; Gene Expression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Immunosuppression Taper (Experimental): Eligible patients who are deemed immune quiescent will undergo sequential withdrawal of immunosuppression medications over a 12-month period from a multi-drug regimen to a Belatacept monotherapy using precision medicine.
  Interventions: Diagnostic Test: Allosure and TruGraf; Other: Immunosuppression Taper
- Multi-Drug Regimen (Other): Eligible patients who are not deemed immune quiescent will continue on a multi-drug regimen.
  Interventions: Diagnostic Test: Allosure and TruGraf

INTERVENTIONS:
Diagnostic Test: Allosure and TruGraf — Precision medicine will be employed to withdraw immunosuppression in kidney transplant recipients.
Other: Immunosuppression Taper — An immunosuppression taper will be employed over a 12-month period for those that are deemed immune quiescent.
  Arms: Immunosuppression Taper

SUMMARY:
The purpose of the study is to provide immunosuppression weaning and/or monitoring for an additional 12-months to evaluate the safety and efficacy of belatacept monotherapy in patients previously enrolled in the clinical trial: "Use of donor derived-cell free DNA (AlloSure) and gene expression profiling (AlloMap Kidney) to facilitate Belatacept monotherapy in kidney transplant patients."

ELIGIBILITY:
Inclusion Criteria:

* Completion of the parent study (STU-2020-1339)
* Able to provide informed consent
* Absence of donor specific antibodies
* Stable renal function (eGFR>40mL/min for 3 months prior to enrollment)

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial
* Significant hepatic impairment
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial
* Proteinuria > 0.5 g/g creatinine on spot urine sample within 3 months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney graft rejection | 12 months after informed consent
  Number of patients with biopsy-proven acute kidney graft rejection
Incidence of facilitation to Belatacept monotherapy | 12 months after the first study visit
  Percentage of subjects successfully weaned to a Belatacept monotherapy

SECONDARY OUTCOMES:
Patient Survival after Immunosuppression Wean | 12 months after informed consent
  Number of patients who died
Kidney Graft Failure after Immunosuppression Wean | 12 months after informed consent
  Number of patients with kidney graft failure. Graft failure is defined as date of patient death or date of re-transplant
Mean change in Estimated Glomerular Filtration Rate (eGFR) after Immunosuppression Wean | 12 months after informed consent
  Estimated glomerular filtration rate (eGFR) in blood will be measured at the beginning of enrollment and the difference will be measured to the end of the study as a measure of change in kidney function.
Incidence of Proteinuria after Immunosuppression Wean | 12 months after informed consent
  Proteinuria will be detected by a semiquantitative method of the protein concentration in urine.
Incidence of de-novo donor specific antibodies (dnDSA) | 12 months after informed consent
  HLA type I and type II in blood will be used to detect the presence of de-novo donor specific antibodies (dnDSA) in those who have started the immunosuppression wean.

CONTACTS AND LOCATIONS:
Overall Officials: David Wojciechowski, DO, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT06336863/Prot_SAP_000.pdf